CLINICAL TRIAL: NCT07245771
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1/2a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Effect on Body Weight of RN3161 as Monotherapy and in Combination With Tirzepatide in Adults With Overweight and Obesity
Brief Title: Phase 1/2a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Effect on Body Weight of RN3161 as Monotherapy and in Combination With Tirzepatide in Adults With Overweight and Obesity
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ikaria Bioscience Pty Ltd (Industry)
Collaborators: Shanghai Rona Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN3161-101
Record Dates: First submitted 2025-09-20; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Obesity &Amp; Overweight
Keywords: obesity; overweight; healthy volunteers
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: randomized to study drug or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- RN3161 (Experimental): Investigational Product
  Interventions: Drug: RN3161
- Placebo Control (Placebo Comparator): placebo control
  Interventions: Drug: Placebo Control
- RN3161 and tirzepatide (Experimental): In Part 3, RN3161 co-administered with tirezepatide
  Interventions: Drug: RN3161; Drug: Tirzepatide
- Placebo and tirzepatide (Active Comparator): In Part 3; Placebo co-administered with tirzepatide
  Interventions: Drug: Placebo Control; Drug: Tirzepatide

INTERVENTIONS:
Drug: RN3161 — Investigational Product
  Arms: RN3161; RN3161 and tirzepatide
Drug: Placebo Control — 0.9% normal saline SC injection
  Arms: Placebo Control; Placebo and tirzepatide
Drug: Tirzepatide — In Part 3; randomized to either RN3161 + tirzepatide or placebo + tirzepatide
  Arms: Placebo and tirzepatide; RN3161 and tirzepatide

SUMMARY:
Study to assess the safety, pharmacokinetics (the amount of study drug or any of its breakdown products in your body) and pharmacodynamics (how the study drug affects your body) of RN3161 alone (healthy volunteers) and RN3161 with tirzepatide (overweight and obese subjects)

ELIGIBILITY:
Inclusion Criteria:

* BMI:

Obesity: BMI ≥ 30 kg/m² for participants with no Asian ancestry and ≥ 27.5 kg/m² for participants with Asian ancestry that has been stable (± 5%) for the previous 3 months (based on participant self-report or available medical records), with or without a weight-related comorbidity (excluding diabetes)

Overweight: BMI 27 to <30 kg/m² for participants with no Asian ancestry and 23.0 to <27.5 kg/m² for participants with Asian ancestry that has been stable (± 5%) for the previous 3 months (based on participant self-report or available medical records), with at least 1 weight-related comorbidity (excluding diabetes)

Weight-related comorbidities include a diagnosis of the following:

* Hypertension: seated BP ≤ 140/90 mm Hg; receiving ≤ 2 stable (≥ 4 weeks) agents limited to ACE inhibitors, angiotensin receptor blockers, calcium channel blockers, or thiazide ≤ 25 mg, or untreated
* Dyslipidemia: stable use of lipid-lowering agents for dyslipidemia (LDL-C < 150 mg/dL, triglycerides < 300 mg/dL)
* Osteoarthritis

Exclusion Criteria:

* self-reported or documented weight gain or loss >5% within 3 months prior to screening
* use of GLP1R agonists within 6 months of screening
* intolerance to GLP-1 medications in the past
* use of non-GLP1R medications for weight loss within 3 months of screening
* HbA1c >6.5%
* diagnosis of significant liver disease
* history of malignancy or anaphylaxis
* use of any siRNA agent in the prior 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 180 Days
  Number of participants with blood pressure changes measured in mmHg
ECG PR interval | 180 days
  Number of participants with change in PR interval measured as milliseconds
Physical Examination | 180 days
  Number of participants with changes seen by physical examination of skin, lymph nodes, eyes, ears, throat, chest, abdomen, musculoskeletal system and nervous system
Blood Chemistry Laboratory | 180 days
  Number of participants with changes in blood levels of sodium, potassium, chloride, calcium magnesium, creatinine, bilirubin, phosphate, AST, ALT, alkaline phosphatase, glucose, albumin, urea in standard units
Adverse Events | 180 days
  Incidence of adverse events reported
Heart Rate | 180 days
  Number of participants with change in heart rate measured in beats per minute
ECG QRS Complex | 180 days
  Number of participants with changes in QRS complex measured in milliseconds
ECG QT interval | 180 days
  Number of participants with change in QT interval measured by Frederica method in milliseconds
Blood Hematology Laboratory | 180 days
  Number of participants with changes in blood hemoglobin, hematocrit, platelets, neutrophils and leukocytes measured in standard units
Blood Coagulation Laboratory | 180 days
  Number of participants with changes in plasma prothrombin time, activated partial thromboplastin time, and international normalized ratio measured in standard units

SECONDARY OUTCOMES:
Plasma and Urine Pharmacokinetics | 180 Days
  plasma and urine levels of RN3161
Presence of ADA | 180 days
  incidence of anti-drug antibodies in the plasma

OTHER OUTCOMES:
Effect of RN3161 on plasma insulin | 180 days
  assess plasma insulin uU/mL
Assess RN3161 effect on plasma LDL | 180 days
  LDL-C in mg/dL
Effect of RN3161 on plasma HDL | 180 days
  HDL in mg/dL
Effect of RN3161 on plasma total cholesterol | 180 days
  total cholesterol in mg/dL
Effect of RN3161 on plasma triglycerides | 180 days
  triglycerides in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Philip Ryan, MD, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The plan will be developed during study conduct.